CLINICAL TRIAL: NCT07277192
Title: HAIC vs. TACE Combined With ICIs and TKIs in Intermediate-to-Advanced HCC: A Multicenter Study on Liver Injury and Survival
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-571
Record Dates: First submitted 2025-11-13; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Hepatecellular Carcinoma; Liver Injury; HAIC(Hepatic Artery Infusion Chemotherapy); TACE(Transcatheter Arterial Chemoembolization)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HAIC-group: HAIC combined with ICIs and TKIs
- TACE-group: TACE combined with ICIs and TKIs

SUMMARY:
The purpose of this study is to compare the liver injury induced by HAIC combined with PD-1/PD-L1 inhibitors and TKIs versus triple therapy with TACE in the treatment of patients with advanced HCC; to compare the efficacy of the two triple therapy regimens in the treatment of patients with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily join this study and sign the informed consent form;
* Aged ≥ 18 years, both male and female;
* Patients with pathologically or clinically confirmed BCLC stage B or C hepatocellular carcinoma (HCC) who were diagnosed between January 1, 2019, and December 31, 2022;
* Receiving treatment with PD-1/PD-L1 inhibitors combined with anti-angiogenic drugs (both PD-1/PD-L1 inhibitors and targeted drugs are only approved post-market medications, including but not limited to those with HCC indications);
* Transarterial chemoembolization (TACE) or hepatic arterial infusion chemotherapy (HAIC) completed within 3 months after the first systemic treatment or within 1 month before the first systemic treatment;
* Having at least one measurable intrahepatic lesion, with intrahepatic lesions being the main tumor burden. (According to RECIST v1.1, the measurable lesion has a spiral CT scan long diameter ≥ 10 mm or enlarged lymph node short diameter ≥ 15 mm).

Exclusion Criteria:

* Pathologically/histologically confirmed cholangiocarcinoma, combined hepatocellular-cholangiocarcinoma, sarcomatoid hepatocellular carcinoma, or fibrolamellar hepatocellular carcinoma;
* Patients with a history of other malignant tumors within the past 3 years or concurrent malignant tumors (except cured basal cell carcinoma of the skin and cervical in situ carcinoma);
* Concomitant use of other antitumor therapeutic agents, such as antitumor traditional Chinese medicines and proprietary Chinese medicines;
* Patients who do not meet the definition of combination therapy;
* Incomplete medical information, such as lack of post-treatment imaging evaluation;
* Patients with immunodeficiency or those who have undergone organ/bone marrow transplantation;
* Patients deemed unsuitable to participate in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intermediate-to-Advanced HCC who received HAIC/TACE combined with PD-1/PD-L1 inhibitors combined with anti-angiogenic drugs (both PD-1/PD-L1 inhibitors and targeted drugs
Sampling Method: Non-Probability Sample
Enrollment: 562 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
alanine aminotransferase(ALT) | Measurements were conducted one week before the first treatment and at regular intervals for up to six months after the intervention, continuing until the occurrence of unacceptable toxicity, withdrawal of consent, or termination of the study by the spon

SECONDARY OUTCOMES:
The median progression free survival time (mPFS) | From date of first dose of study drug to the date of first documentation of disease progression or death, whichever occurs first (up to approximately 3 years)
  The progression free survival time defined as the time from the first study dose date to the date of first documentation of disease progression as assessed by RECIST 1.1
The median overall survival time (mOS) | From date of first dose of study drug to the date of first documentation of disease progression or death, whichever occurs first (up to approximately 3 years)
  Overall survival rate is measured from the start date of the Treatment Phase (date of first study dose) until date of death from any cause. Participants who are lost to follow-up and the participants who are alive at the date of data cutoff will be censored at the date the participant was last known alive or the cut-off date, whichever comes early.
Objective response rate (ORR) | From date of first dose of study drug until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to approximately 3 years)
The disease control rate (DCR) | From date of first dose of study drug until disease progression, stable disease, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to approximately 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhang Chen, Study Director — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No